CLINICAL TRIAL: NCT00574327
Title: A Prospective Study To Define The Role Of Various Factors In Development And Progression Of Gastroesophageal Reflux Disease (GERD) And Barrett's Esophagus And The Creation Of A Registry.
Brief Title: Progression of Gastroesophageal Reflux Disease and Barrett's Esophagus and the Creation of a Barrett's Registry
Status: Recruiting | Type: Observational
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: PS0035
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Barrett's Esophagus; Gastroesophageal Reflux Disease; Esophageal Adenocarcinoma
Keywords: Role; Registry; Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples from participating patients will be collected and frozen for measurements of insulin, glucose, lipid panel, CRP and adiponectin levels. Biopsies obtained from esophagus during endoscopy and blood samples will be frozen for future biomarker and cDNA microarray studies and histochemistry.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A- Barrett's Esophagus subjects: Patients with documented Barrett's Esophagus with or without dysplasia (LGD or HGD) that will undergo surveillance endoscopies dictated by the grade of dysplasia.
- B- gastroesophageal reflux subjects: Patients undergoing endoscopy for evaluation of GERD symptoms.
- C-subjects without BE or GERD: The control group would include patients undergoing upper endoscopy for reasons other than stated above, such as evaluation of iron deficiency anemia, weight loss, positive fecal occult blood, etc.

SUMMARY:
The purpose of this study is to determine or evaluate the risk factors such as smoking, family history etc. that cause esophageal cancer and to determine the genetic changes that lead to esophageal cancer. The investigators hypothesis is that systematic collection of data on the natural history of GERD and BE patients and risk factors for development of BE in patients with chronic GERD and progression of BE to dysplasia and adenocarcinoma will provide useful information to develop a decision model for risk stratification and risk reduction strategies in these patients.

As of March 17, 2011, 585 patients have consented at the Kansas City VA Medical Center.

DETAILED DESCRIPTION:
Symptoms of gastroesophageal reflux are common. It affects at least 40% of the adult American population and 40 million American adults experience reflux symptoms on a regular basis. Gastroesophageal reflux disease (GERD) typically affects Caucasians and older males. It is a significant risk factor for development of Barrett's esophagus (BE) and esophageal adenocarcinoma. Approximately 10-15% of patients with chronic GERD are diagnosed with BE, a premalignant lesion for esophageal adenocarcinoma. Adenocarcinoma of the esophagus continues to be the most rapidly increasing incidence cancer in the United States. Based on studies evaluating screening/surveillance strategies, it is clear that it is imperative to identify risk factors that would target those patients with gastroesophageal reflux disease (GERD) and BE that may benefit from screening and surveillance strategies, yet also be practical and cost-effective. A better understanding of the events surrounding the development of BE in patients with chronic GERD, development of dysplastic changes in patients with BE and progression of BE to adenocarcinoma may ultimately help in identifying those patients at increased risk. Thus, our hypothesis is that systematic collection of data on the natural history of GERD and BE patients and risk factors for development of BE in patients with chronic GERD and progression of BE to dysplasia and adenocarcinoma will provide useful information to develop a decision model for risk stratification and risk reduction strategies in these patients. This model will be a useful tool leading to a reduction in overall health care costs.

The study will be conducted at the Kansas City Department of Veterans Affairs Medical Center. This is a prospective cohort study designed to analyze the epidemiologic and genetic factors relevant to development of BE in patients with GERD and its subsequent progression to dysplasia and adenocarcinoma. 1) The consenting patients as well as controls (2:1 ratio) will be asked to fill validated questionnaire on severity of GERD and food frequency. Data regarding medications, family history and social history will also be collected. 2) The endoscopy and pathology reports will be browsed for length of Barrett's esophagus confirmed by histology, length of hiatal hernia and presence of helicobacter pylori. 3) Serum samples from participating patients will be collected and frozen for measurements of insulin, glucose, lipid panel, CRP and adiponectin levels. Biopsies obtained from esophagus during endoscopy and blood samples would be frozen for future biomarker and cDNA microarray studies and histochemistry.

Approximately10-20% of the adult population has GERD and 0.5 to 2% of the adult population (1-4 million individuals) is estimated to have BE and it is a known precursor to esophageal adenocarcinoma. However, we are not yet able to reliably identify those individuals with GERD that are at risk for developing BE and with BE who are at high risk for progressing to esophageal adenocarcinoma. The identification of risk factors as the ultimate goal of this study will enable us to better identify the high-risk patients and provide early intervention and therapeutic strategies in a cost-effective manner.

ELIGIBILITY:
All patients must be eligible for care that the Kansas City VA Hospital where this study was approved for enrollment.

Inclusion Criteria:

* Kansas City VA Patients with confirmed BE with and without dysplasia and patients with reflux disease (patients/cases); patients with other indicators for endoscopy such as anemia, weight loss, diarrhea, but without GERD and PE (controls).

Exclusion Criteria:

* Patients with uncontrolled significant comorbidities such as cardiovascular, pulmonary, renal, hepatic or metabolic diseases.
* Presence of anticoagulation that would increase risk from biopsies
* Patients unable to provide history
* Patients with dyspepsia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients must be eligible for care at the Kansas City VA Medical Center. Those presenting to the Kansas City VA endoscopy laboratory for their "standard BE surveillance" endoscopy. Patients with a history of BE will be identified and contacted from the existing databank. Patients with newly diagnosed BE in the endoscopy laboratory after their procedure is completed and biopsy results are available. Patients undergoing upper endoscopy for evaluation of GERD symptoms. Control group of patients undergoing upper endoscopy for any reason other than the ones stated above.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2006-01; Primary Completion 2028-10 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
The goal of this study is to follow GERD and BE pts prospectively for development of dysplasia and adenocarcinoma, to identify factors responsible for progression of GERD to BE to dysplasia and adenocarcinoma. | 5 plus years

SECONDARY OUTCOMES:
The secondary goal is to create a tissue and serum repository for future biomarker studies. | 5 plus years

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Department of Veterans Affairs Medical Center of Kansas City
Locations (1):
- Department of Veterans Affairs Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Background] Sampliner RE; Practice Parameters Committee of the American College of Gastroenterology. Updated guidelines for the diagnosis, surveillance, and therapy of Barrett's esophagus. Am J Gastroenterol. 2002 Aug;97(8):1888-95. doi: 10.1111/j.1572-0241.2002.05910.x. No abstract available. PMID 12190150
- [Background] Haggitt RC. Barrett's esophagus, dysplasia, and adenocarcinoma. Hum Pathol. 1994 Oct;25(10):982-93. doi: 10.1016/0046-8177(94)90057-4. PMID 7927321
- [Background] Reid BJ. Barrett's esophagus and esophageal adenocarcinoma. Gastroenterol Clin North Am. 1991 Dec;20(4):817-34. PMID 1787015
- [Background] van Sandick JW, van Lanschot JJ, Kuiken BW, Tytgat GN, Offerhaus GJ, Obertop H. Impact of endoscopic biopsy surveillance of Barrett's oesophagus on pathological stage and clinical outcome of Barrett's carcinoma. Gut. 1998 Aug;43(2):216-22. doi: 10.1136/gut.43.2.216. PMID 10189847
- [Background] Gudlaugsdottir S, van Blankenstein M, Dees J, Wilson JH. A majority of patients with Barrett's oesophagus are unlikely to benefit from endoscopic cancer surveillance. Eur J Gastroenterol Hepatol. 2001 Jun;13(6):639-45. doi: 10.1097/00042737-200106000-00005. PMID 11434588
- [Background] van der Burgh A, Dees J, Hop WC, van Blankenstein M. Oesophageal cancer is an uncommon cause of death in patients with Barrett's oesophagus. Gut. 1996 Jul;39(1):5-8. doi: 10.1136/gut.39.1.5. PMID 8881798
- [Background] O'Connor JB, Falk GW, Richter JE. The incidence of adenocarcinoma and dysplasia in Barrett's esophagus: report on the Cleveland Clinic Barrett's Esophagus Registry. Am J Gastroenterol. 1999 Aug;94(8):2037-42. doi: 10.1111/j.1572-0241.1999.01275.x. PMID 10445525
- [Background] Wong A, Fitzgerald RC. Epidemiologic risk factors for Barrett's esophagus and associated adenocarcinoma. Clin Gastroenterol Hepatol. 2005 Jan;3(1):1-10. doi: 10.1016/s1542-3565(04)00602-0. PMID 15645398
- [Background] Shirvani VN, Ouatu-Lascar R, Kaur BS, Omary MB, Triadafilopoulos G. Cyclooxygenase 2 expression in Barrett's esophagus and adenocarcinoma: Ex vivo induction by bile salts and acid exposure. Gastroenterology. 2000 Mar;118(3):487-96. doi: 10.1016/s0016-5085(00)70254-x. PMID 10702199
- [Background] Wilson KT, Fu S, Ramanujam KS, Meltzer SJ. Increased expression of inducible nitric oxide synthase and cyclooxygenase-2 in Barrett's esophagus and associated adenocarcinomas. Cancer Res. 1998 Jul 15;58(14):2929-34. PMID 9679948
- [Background] Rabinovitch PS, Longton G, Blount PL, Levine DS, Reid BJ. Predictors of progression in Barrett's esophagus III: baseline flow cytometric variables. Am J Gastroenterol. 2001 Nov;96(11):3071-83. doi: 10.1111/j.1572-0241.2001.05261.x. PMID 11721752
- [Background] Reid BJ, Levine DS, Longton G, Blount PL, Rabinovitch PS. Predictors of progression to cancer in Barrett's esophagus: baseline histology and flow cytometry identify low- and high-risk patient subsets. Am J Gastroenterol. 2000 Jul;95(7):1669-76. doi: 10.1111/j.1572-0241.2000.02196.x. PMID 10925966
- [Background] Cameron AJ, Lomboy CT. Barrett's esophagus: age, prevalence, and extent of columnar epithelium. Gastroenterology. 1992 Oct;103(4):1241-5. doi: 10.1016/0016-5085(92)91510-b. PMID 1397881
- [Background] El-Serag HB, Petersen NJ, Carter J, Graham DY, Richardson P, Genta RM, Rabeneck L. Gastroesophageal reflux among different racial groups in the United States. Gastroenterology. 2004 Jun;126(7):1692-9. doi: 10.1053/j.gastro.2004.03.077. PMID 15188164
- [Background] Younes M, Henson DE, Ertan A, Miller CC. Incidence and survival trends of esophageal carcinoma in the United States: racial and gender differences by histological type. Scand J Gastroenterol. 2002 Dec;37(12):1359-65. doi: 10.1080/003655202762671215. PMID 12523583
- [Background] Lagergren J, Bergstrom R, Lindgren A, Nyren O. Symptomatic gastroesophageal reflux as a risk factor for esophageal adenocarcinoma. N Engl J Med. 1999 Mar 18;340(11):825-31. doi: 10.1056/NEJM199903183401101. PMID 10080844
- [Background] Gray MR, Donnelly RJ, Kingsnorth AN. The role of smoking and alcohol in metaplasia and cancer risk in Barrett's columnar lined oesophagus. Gut. 1993 Jun;34(6):727-31. doi: 10.1136/gut.34.6.727. PMID 8314502
- [Background] Vaughan TL, Davis S, Kristal A, Thomas DB. Obesity, alcohol, and tobacco as risk factors for cancers of the esophagus and gastric cardia: adenocarcinoma versus squamous cell carcinoma. Cancer Epidemiol Biomarkers Prev. 1995 Mar;4(2):85-92. PMID 7742727
- [Background] Terry P, Lagergren J, Hansen H, Wolk A, Nyren O. Fruit and vegetable consumption in the prevention of oesophageal and cardia cancers. Eur J Cancer Prev. 2001 Aug;10(4):365-9. doi: 10.1097/00008469-200108000-00010. PMID 11535879
- [Background] Chow WH, Blot WJ, Vaughan TL, Risch HA, Gammon MD, Stanford JL, Dubrow R, Schoenberg JB, Mayne ST, Farrow DC, Ahsan H, West AB, Rotterdam H, Niwa S, Fraumeni JF Jr. Body mass index and risk of adenocarcinomas of the esophagus and gastric cardia. J Natl Cancer Inst. 1998 Jan 21;90(2):150-5. doi: 10.1093/jnci/90.2.150. PMID 9450576
- [Background] Moe GL, Kristal AR, Levine DS, Vaughan TL, Reid BJ. Waist-to-hip ratio, weight gain, and dietary and serum selenium are associated with DNA content flow cytometry in Barrett's esophagus. Nutr Cancer. 2000;36(1):7-13. doi: 10.1207/S15327914NC3601_2. PMID 10798210
- [Background] Romero Y, Cameron AJ, Locke GR 3rd, Schaid DJ, Slezak JM, Branch CD, Melton LJ 3rd. Familial aggregation of gastroesophageal reflux in patients with Barrett's esophagus and esophageal adenocarcinoma. Gastroenterology. 1997 Nov;113(5):1449-56. doi: 10.1053/gast.1997.v113.pm9352846.
- [Background] Lagergren J, Bergstrom R, Adami HO, Nyren O. Association between medications that relax the lower esophageal sphincter and risk for esophageal adenocarcinoma. Ann Intern Med. 2000 Aug 1;133(3):165-75. doi: 10.7326/0003-4819-133-3-200008010-00007. PMID 10906830
- [Background] El-Serag HB, Aguirre TV, Davis S, Kuebeler M, Bhattacharyya A, Sampliner RE. Proton pump inhibitors are associated with reduced incidence of dysplasia in Barrett's esophagus. Am J Gastroenterol. 2004 Oct;99(10):1877-83. doi: 10.1111/j.1572-0241.2004.30228.x. PMID 15447744
- [Background] Corley DA, Kerlikowske K, Verma R, Buffler P. Protective association of aspirin/NSAIDs and esophageal cancer: a systematic review and meta-analysis. Gastroenterology. 2003 Jan;124(1):47-56. doi: 10.1053/gast.2003.50008. PMID 12512029
- [Background] Freedman J, Ye W, Naslund E, Lagergren J. Association between cholecystectomy and adenocarcinoma of the esophagus. Gastroenterology. 2001 Sep;121(3):548-53. doi: 10.1053/gast.2001.27217. PMID 11522738
- [Background] McDonald ML, Trastek VF, Allen MS, Deschamps C, Pairolero PC, Pairolero PC. Barretts's esophagus: does an antireflux procedure reduce the need for endoscopic surveillance? J Thorac Cardiovasc Surg. 1996 Jun;111(6):1135-8; discussion 1139-40. doi: 10.1016/s0022-5223(96)70214-3. PMID 8642813
- [Background] Trujillo ME, Scherer PE. Adiponectin--journey from an adipocyte secretory protein to biomarker of the metabolic syndrome. J Intern Med. 2005 Feb;257(2):167-75. doi: 10.1111/j.1365-2796.2004.01426.x. PMID 15656875
- [Background] Weston AP, Sharma P, Mathur S, Banerjee S, Jafri AK, Cherian R, McGregor D, Hassanein RS, Hall M. Risk stratification of Barrett's esophagus: updated prospective multivariate analysis. Am J Gastroenterol. 2004 Sep;99(9):1657-66. doi: 10.1111/j.1572-0241.2004.30426.x. PMID 15330898
- [Background] Weston AP, Badr AS, Topalovski M, Cherian R, Dixon A, Hassanein RS. Prospective evaluation of the prevalence of gastric Helicobacter pylori infection in patients with GERD, Barrett's esophagus, Barrett's dysplasia, and Barrett's adenocarcinoma. Am J Gastroenterol. 2000 Feb;95(2):387-94. doi: 10.1111/j.1572-0241.2000.01758.x. PMID 10685740
- [Background] Kan T, Shimada Y, Sato F, Maeda M, Kawabe A, Kaganoi J, Itami A, Yamasaki S, Imamura M. Gene expression profiling in human esophageal cancers using cDNA microarray. Biochem Biophys Res Commun. 2001 Aug 31;286(4):792-801. doi: 10.1006/bbrc.2001.5400. PMID 11520067
- [Background] Souza RF, Morales CP, Spechler SJ. Review article: a conceptual approach to understanding the molecular mechanisms of cancer development in Barrett's oesophagus. Aliment Pharmacol Ther. 2001 Aug;15(8):1087-100. doi: 10.1046/j.1365-2036.2001.01046.x. PMID 11472311
- [Derived] Bansal A, Lee IH, Hong X, Anand V, Mathur SC, Gaddam S, Rastogi A, Wani SB, Gupta N, Visvanathan M, Sharma P, Christenson LK. Feasibility of mcroRNAs as biomarkers for Barrett's Esophagus progression: a pilot cross-sectional, phase 2 biomarker study. Am J Gastroenterol. 2011 Jun;106(6):1055-63. doi: 10.1038/ajg.2011.37. Epub 2011 Mar 15. PMID 21407181